CLINICAL TRIAL: NCT00661219
Title: A Randomized Double-blind Multi-center Parallel Group Three Month Study to Compare the Tolerability and Efficacy of Flexible Dose Vardenafil Versus Placebo in Men With Depression and Erectile Dysfunction.
Brief Title: Depression Related Improvement With Vardenafil for Erectile Response
Acronym: DRIVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10621
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction; Depression
MeSH Terms: conditions — Erectile Dysfunction; Depression | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — BAY 38-9456 (vardenafil) will be supplied as 5 mg tablets, 10 mg tablets, and 20 mg tablets.
  Arms: Arm 1
Drug: Placebo — Identical placebo will be matched for each vardenafil dosage form and will be indistinguishable from active treatment.
  Arms: Arm 2

SUMMARY:
The study will last three months. During the first month of treatment the subject will receive either 10 mg vardenafil or placebo. After 1 month of treatment the doctor, can choose to increase the dosage from 10 mg to 20 mg or decrease the dosage to 5 mg. The doctor will again evaluate, after 2 months of treatment if the subject wants to increase the dosage from 10 mg to 20 mg or, if already done, to continue with the dosage of 20 mg or decrease to 10 mg or 5 mg. It will not be possible after this point to increase or decrease the dosage for the rest of the study. The subject will be asked to attend the clinic on four separate occasions over a period of 3 months. Every visit will last about 1 hour. At the first visit the doctor will ask the subject about their medical history, and the subject will be given a medical examination (including your heart rate, blood pressure and weight). The medical examination will also include an ECG. The subject will be asked to provide a blood and urine sample, which will be analysed and screened for drugs of potential abuse (e.g.cocaine, narcotics, sedatives, hypnotics). The subject will then be asked to fill in a questionnaire about their mood and feelings. The subject qualifies, they will have an interview with a trained mental health care provider who will assess their level of depression. At the end of the visit, the doctor will provide the subject with a diary in which they must record details about their attempts at sexual activity during the next 4 weeks. The subject will be asked to make at least 4 attempts at sexual intercourse on 4 separate days and to record the attempts in the diaries. After 4 weeks the subject will return to the clinic. They will be asked to fill in different questionnaires about their sexuality, mood and feelings, general quality of life, self-esteem and sexual activity in the last 4 weeks. Two additional blood and urine samples will be collected. An interview with the trained mental health care provider who will re-assess their level of depression. At this visit all information collected so far will be assessed and the doctor will check to see if the requirements to enter the treatment period are fulfilled. The subject may be excluded from further participation in the study, for example due to results of the blood analysis or if your level of depression did not meet the criteria for the study. If the subject is able to participate to the study they will be given the study drug. At each visit, adverse events will be discussed and whether there is any change in medicine. Vital signs and ECG will be obtained at visit one, two, five and/or Premature Termination. At every visit the subject will receive a diary in which they must record details about their attempts at sexual activity during the period between each visit and the number of tablets taken. Subjects will also be asked to fill in different questionnaires about their sexuality, mood and feelings, self-esteem and sexual activity. Subjects will also be contacted by telephone, at 2, 6 and 10 weeks after starting the study medication, 24 hours after the last dose of study medication. The doctor will give the study drug on 3 occasions. Should the subject or doctor prematurely stop trial participation the subject will be required to return to the clinic for a physical examination, vital signs and have blood samples and ECG obtained. They will also be asked to fill in different questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction for more than 6 months according to the NIH Consensus statement (the inability to attain and maintain erection of the penis sufficient to permit satisfactory sexual intercourse).
* Stable, heterosexual relationship for more than 6 months.
* Diagnosis of mild Major Depressive Disorder using a structured interview (SCID-1 or MINI), according to DSM-IV criteria. Before randomization, a psychiatrist must interview the subject at Visit 2 to validate both the diagnosis of MDD and the subject's continuation in the study without the need for anti-depressant medication or psychotherapy).
* Patients must score greater than 13 on the CES-D at Visit 1.
* Patients must score between 11 and 17 on the 17-item HAM-D at Visit 1 and Visit 2.
* The patient must make at least four attempts at sexual intercourse on four separate days during the untreated baseline period
* At least 50% of the attempts of sexual intercourse during the untreated baseline period have to be unsuccessful

Exclusion Criteria:

Previous or Current Medical Conditions

* Any unstable medical condition or substance abuse disorder that, in the opinion of the Investigator, is likely to affect the patient's ability to complete the study or precludes the patient's participation in the study.
* Patients who score > 0 on item #3 on the HAM-D17 or men who, in the investigator's judgement, pose a current serious suicidal or homicidal risk or have made a suicide attempt within the past 12 months.
* Men with a current (or within 6 months prior to screening) Axis 1 disorder other than MDD (major depressive disorder). Patients with a history, or who currently meet the DSM-IV criteria, of Bipolar Disorder, Schizophrenia, Schizoaffective Disorder, Delusional (Paranoid) Disorder, Panic Disorder, Post-Traumatic Stress Disorder. Patients with a Personality Disorder are excluded if, in the investigator's opinion, it will interfere with the conduct of the trial.
* Retinitis pigmentosa.
* Unstable angina pectoris.
* History of radical prostatectomy.
* History of myocardial infarction, stroke, electrocardiographic ischemia (except stable angina), or life-threatening arrhythmia within the prior 6 months.

Abnormal Laboratory Values

* AST or ALT > 3 times the upper limit of normal Concomitant Medications
* Patients who are taking nitrates or nitric oxide donors (e.g., molsidomine, minoxidil). Topical minoxidil is permitted.
* Patients who are taking androgens (e.g., testosterone) or anti-androgens.
* Patients taking trazodone, or any other anti-depressant including monoamine oxidase inhibitors, St. John's Wort, SSRIs or tricyclic anti-depressants are excluded, or use of these medications in the last 2 weeks before Visit 1. Fluoxetine is excluded in the last 4 weeks before Visit 1.
* Patients who are taking the following potent inhibitors of cytochrome P 450 3A4: the HIV protease inhibitors ritonavir and indinavir, erythromycin or the anti-mycotic agents itraconazole and ketoconazole (topical forms are allowed).
* Subjects who are taking alpha-blockers.
* Use of any therapy for erectile dysfunction within seven days of Visit 1 and during the trial.
* Patients who require, or are likely to require, treatment with psychotherapy or psychotropic drugs during the course of the study. Men receiving formal individual psychotherapy for depression currently or in the 12 weeks prior to screening visit.

Abnormal Laboratory Values

* Patients who have a serum total testosterone level >10% below the lower limit of normal (according to the range specified by the responsible laboratory).

Other Exclusions

* Patients whose urine screen for substances of abuse is positive.
* Patients unwilling to refrain from consuming grapefruit juice or products containing grapefruit juice with study medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2002-12; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variables are the change from baseline in the IIEF-EF domain score and the change from baseline in the HAM-D17 total score. | 12 weeks and LOCF

SECONDARY OUTCOMES:
Patient Diary questions of treatment compared to placebo. | 4, 8, and 12 weeks
Global assessment question (GAQ) of treatment compared to placebo. | 12 weeks
The scores for the IIEF questionnaire. | 12 weeks
Responses on the Center for Epidemiologic Studies Depression Scale (CES-D). | 12 weeks
Responses on the Rosenberg Self Esteem Scale. | 12 weeks
Responses on the Clinical Global Impressions scale, Items 1 and 2. | 12 weeks
Reliability in early responders. | 12 weeks
Other IIEF domain scores than EF domain score at 12 weeks. | 12 weeks
Safety assessment | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (44):
- United States (14):
  - Huntsville, Alabama
  - Anchorage, Alaska
  - Beverly Hills, California
  - Irvine, California
  - La Mesa, California
  - San Diego, California
  - Aventura, Florida
  - Atlanta, Georgia
  - Boston, Massachusetts
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Durham, North Carolina
  - Charlottesville, Virginia
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Markham, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Hull, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Sherbrooke, Quebec
- France (6):
  - Lille
  - Lyon
  - Marseille
  - Nantes
  - Nice
  - Paris
- Italy (8):
  - Bari
  - Florence
  - Milan
  - Modena
  - Napoli
  - Padua
  - Pisa
  - Roma
- Spain (5):
  - Barcelona, Barcelona
  - Galdakao, Bizkaia
  - Madrid, Madrid
  - Seville, Sevilla
  - Zaragoza, Zaragoza